CLINICAL TRIAL: NCT01122680
Title: A Phase II Randomised, Double-blind, Placebo-controlled, Incomplete Crossover Trial With 4-week Treatment Periods to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution (Doses of 1.25 µg, 2.5 µg and 5 µg) Delivered Via Respimat® Inhaler Once Daily in the Evening in Adolescents (12 to 17 Yrs Old) With Moderate Persistent Asthma
Brief Title: Efficacy and Safety of 3 Doses of Tiotropium Compared to Placebo in Adolescents (12 to 17 Yrs) With Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.424; 2009-017745-55 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (4):
- Treatment A (Experimental): patients inhale 2 puffs (dose of 1.25 mcg) once daily in the evening via Respimat inhaler
  Interventions: Drug: Tiotropium bromide
- Treatment C (Experimental): patients inhale 2 puffs (dose of 5 mcg) once daily in the evening via Respimat inhaler
  Interventions: Drug: tiotropium bromide
- Placebo (Placebo Comparator): patients inhale 2 puffs of placebo matching tiotropium once daily in the evening via Respimat inhaler
  Interventions: Drug: Placebo
- Treatment B (Experimental): patients inhale 2 puffs (dose of 2.5 mcg) once daily in the evening via Respimat inhaler
  Interventions: Drug: tiotropium bromide

INTERVENTIONS:
Drug: Tiotropium bromide — inhalation solution, dose of 1.25 mcg (2 puffs of 0.625 mcg)
  Arms: Treatment A
Drug: tiotropium bromide — inhalation solution, dose of 2.5 mcg (2 puffs of 1.25 mcg)
  Arms: Treatment B
Drug: tiotropium bromide — inhalation solution, dose of 5 mcg (2 puffs of 2.5 mcg)
  Arms: Treatment C
Drug: Placebo — placebo inhalation solution
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to evaluate the efficacy and safety of tiotropium 1.25 mcg (2 actuations of 0.625 mcg), tiotropium 2.5 mcg (2 actuations of 1.25 mcg) and tiotropium 5 mcg (2 actuations of 2.5 mcg) once daily in the evening delivered by the Respimat inhaler in adolescents (12 to 17 yrs) with moderate persistent asthma, compared to placebo and on top of maintenance therapy with an inhaled corticosteroid controller medication. It is a randomised, double-blind, placebo-controlled Phase II trial with incomplete cross-over design. Patients need to be still symptomatic, i. e. not fully controlled with their maintenance treatment.

ELIGIBILITY:
Inclusion criteria:

1. All patients and legally accepted caregiver(s) must sign and date an Informed Consent form consistent with Good Clinical Practice (GCP) guidelines of the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and local legislation prior to participation in the trial.
2. Male or female patients between 12 and 17 years of age.
3. All patients must have at least a 3 months history of asthma and fulfill the diagnostic criteria of moderate persistent asthma, according to the current Global Initiative for Asthma (GINA) guidelines at the time of enrolment into the trial.
4. All patients must have been on maintenance treatment with inhaled corticosteroids at a stable medium dose for at least 4 weeks before Visit 1.
5. All patients must be symptomatic (partly controlled) at Visit 1 (screening) and prior to randomisation at Visit 2 as defined by an Asthma Control Questionnaire (ACQ) mean score of equal or above 1.5.
6. All patients must have a pre-bronchodilator FEV1 above 60% and less than or equal 90% of predicted normal at Visit 1. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator) as compared to Visit 2 (pre-dose) must be within ± 30%.
7. All patients must have an increase in FEV1 of equal or above 12% and 200 mL 15 min. after 400 mcg salbutamol (albuterol) at Visit 1. If patients in the lower age range (e.g., 12 to 14 year olds) exhibit a very small total lung volume, positive reversibility testing might be based solely on the relative (12%) post-bronchodilator response.
8. All patients should be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment.
9. Patients should be able to use the Respimat® inhaler correctly.
10. Patients must be able to perform all trial related procedures including technically acceptable spirometric manoeuvres, according to American Thoracic Society (ATS) standards and the use of the electronic diary/peak flow meter.

Exclusion criteria:

1. Patients with a significant disease other than asthma.
2. Patients with a history of congenital or acquired heart disease, and/or have been hospitalised for cardiac syncope or failure during the past year.
3. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention (e. g. pacemaker implantation) or a change in drug therapy within the past year.
4. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years.
5. Patients with lung diseases other than asthma, e.g. cystic fibrosis (CF). In case of ex-premature infants, a history of significant bronchopulmonary dysplasia (BPD) will be regarded as exclusion criterion
6. Patients with significant alcohol or drug abuse within the past two years.
7. Patients with known hypersensitivity to anticholinergic drugs, benzalkonium chloride (BAC), ethylenediaminetetraacetic acid (EDTA) or any other components of the tiotropium inhalation solution.
8. Pregnant or nursing adolescent female patients, including female patients with a positive Beta HCG (serum pregnancy) testing at screening (visit 1).
9. Sexually active female patients of child-bearing potential not using a highly effective method of birth control.
10. Patients with a known narrow-angle glaucoma, or any other disease where anticholinergic treatment is contraindicated.
11. Patients with renal impairment, as defined by a creatinine clearance less than 50 mL/min/1.73 m2 body surface area (BSA) as calculated by Schwartz Formula.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- United States (5):
  - 205.424.01002 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 205.424.01006 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 205.424.01007 Boehringer Ingelheim Investigational Site, Warrensburg, Missouri
  - 205.424.01004 Boehringer Ingelheim Investigational Site, Boys Town, Nebraska
  - 205.424.01001 Boehringer Ingelheim Investigational Site, Canton, Ohio
- Germany (3):
  - 205.424.49007 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.424.49004 Boehringer Ingelheim Investigational Site, Rosenheim
  - 205.424.49002 Boehringer Ingelheim Investigational Site, Wesel
- Latvia (5):
  - 205.424.37104 Boehringer Ingelheim Investigational Site, Balvi
  - 205.424.37103 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.424.37105 Boehringer Ingelheim Investigational Site, Rēzekne
  - 205.424.37101 Boehringer Ingelheim Investigational Site, Riga
  - 205.424.37102 Boehringer Ingelheim Investigational Site, Riga
- Lithuania (3):
  - 205.424.37001 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.424.37003 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.424.37004 Boehringer Ingelheim Investigational Site, Vilnius
- Slovenia (3):
  - 205.424.38604 Boehringer Ingelheim Investigational Site, Kamnik
  - 205.424.38605 Boehringer Ingelheim Investigational Site, Ljubljana
  - 205.424.38602 Boehringer Ingelheim Investigational Site, Maribor

REFERENCES:
- [Derived] Vogelberg C, Engel M, Moroni-Zentgraf P, Leonaviciute-Klimantaviciene M, Sigmund R, Downie J, Nething K, Vevere V, Vandewalker M. Tiotropium in asthmatic adolescents symptomatic despite inhaled corticosteroids: a randomised dose-ranging study. Respir Med. 2014 Sep;108(9):1268-76. doi: 10.1016/j.rmed.2014.06.011. Epub 2014 Jul 17. PMID 25081651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this incomplete crossover design, 105 patients were randomised to one of four sequences (in general terms, ABC, BDA, CAD or DCB). Whilst there were 4 possible treatments, A, B, C and D, each patient would receive a maximum of 3 different treatments. Hence, approximately 75 patients would receive each of A, B, C and D at any timepoint.
Groups:
- Tio R5/Placebo/Tio R1.25: Patients treated with Tiotropium 5 mcg in Phase I, with a matching Placebo in Phase II and with Tiotropium 1.25 mcg in Phase III. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off-treatment periods) between treatments.
- Tio R1.25/Tio R5/Tio R2.5: Patients treated with Tiotropium 1.25 mcg in Phase I, with Tiotropium 5 mcg in Phase II and with Tiotropium 2.5 mcg in Phase III. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off-treatment periods) between treatments.
- Placebo/Tio R2.5/Tio R5: Patients treated with a matching Placebo in Phase I, with Tiotropium 2.5 mcg in Phase II and with Tiotropium 5 mcg in Phase III. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off-treatment periods) between treatments.
- Tio R2.5/Tio R1.25/Placebo: Patients treated with Tiotropium 2.5 mcg in Phase I, with Tiotropium 1.25 mcg in Phase II and with a matching Placebo in Phase III. All products were administered once daily (QD) in the evening, delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication. No washouts (off-treatment periods) between treatments.
Period: Period 1 (4 Weeks)
Arm/Group | Tio R5/Placebo/Tio R1.25 | Tio R1.25/Tio R5/Tio R2.5 | Placebo/Tio R2.5/Tio R5 | Tio R2.5/Tio R1.25/Placebo
Started | 29 (Entered this study period.) | 26 (Entered this study period.) | 26 (Entered this study period.) | 24 (Entered this study period.)
Completed | 26 (Completed treatment in this crossover period.) | 25 (Completed treatment in this crossover period.) | 26 (Completed treatment in this crossover period.) | 24 (Completed treatment in this crossover period.)
Not Completed | 3 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0
Period: Period 2 (4 Weeks)
Arm/Group | Tio R5/Placebo/Tio R1.25 | Tio R1.25/Tio R5/Tio R2.5 | Placebo/Tio R2.5/Tio R5 | Tio R2.5/Tio R1.25/Placebo
Started | 26 (Entered this study period.) | 25 (Entered this study period.) | 26 (Entered this study period.) | 24 (Entered this study period.)
Completed | 25 (Completed treatment in this crossover period.) | 25 (Completed treatment in this crossover period.) | 26 (Completed treatment in this crossover period.) | 23 (Completed treatment in this crossover period.)
Not Completed | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0 | 0
Period: Period 3 (4 Weeks)
Arm/Group | Tio R5/Placebo/Tio R1.25 | Tio R1.25/Tio R5/Tio R2.5 | Placebo/Tio R2.5/Tio R5 | Tio R2.5/Tio R1.25/Placebo
Started | 25 (Entered this study period.) | 25 (Entered this study period.) | 26 (Entered this study period.) | 23 (Entered this study period.)
Completed | 24 (Completed treatment in this crossover period.) | 24 (Completed treatment in this crossover period.) | 26 (Completed treatment in this crossover period.) | 23 (Completed treatment in this crossover period.)
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total.: Total number of patients randomised and treated at all in the study.
Arm/Group | Total.
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.0 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 67
Forced expiratory volume in 1s (FEV1) [Mean (Standard Deviation); unit: Litre] | 2.742 (0.697)

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume (FEV1) Peak (0-3h) Response
Description: The FEV1 peak (0-3h) response is determined at the end of the 4 week treatment period. This is the difference between the maximum FEV1 measured within the first 3 hours post dosing and the FEV1 baseline measurement. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: The Full analysis set (FAS) is defined as patients randomised, treated, with baseline data and at least one on-treatment efficacy measurement after 4 weeks on treatment within a period. This patient set is therefore FAS reduced to patients with non-missing FEV1 data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Groups:
- Placebo: Placebo once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R1.25: Tiotropium 1.25 microgram once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R2.5: Tiotropium 2.5 microgram once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
- Tio R5: Tiotropium 5 microgram once daily (QD) in the evening delivered by the Respimat® inhaler, on top on maintenance therapy with an inhaled corticosteroid controller medication.
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre | 0.489 (0.047) | 0.556 (0.047) | 0.546 (0.047) | 0.602 (0.046)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Tio R5 minus Placebo; Test type: Superiority or Other; p = 0.0043, Mixed model repeated measures (MMRM) — First step of closed testing procedure, where the active treatments are compared to placebo. If this statisical test significant at the 0.05 alpha level then proceed to comparison of the next lower dose to placebo; This MMRM model includes treatment, period and baseline as fixed effects, and patient as a random effect; Mean Difference (Final Values) = 0.113, 95% CI [0.036 to 0.190], Standard Error of Mean 0.039
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Tio R2.5 minus Placebo; Test type: Superiority or Other; p = 0.1484, Mixed effect repeated measures (MMRM) — Second step of closed testing procedure. If this statisical test significant at the 0.05 alpha level then proceed to comparison of the next lower dose to placebo; This MMRM model includes treatment, period and baseline as fixed effects, and patient as a random effect; Mean Difference (Final Values) = 0.057, 95% CI [-0.021 to 0.135], Standard Error of Mean 0.039
Statistical Analysis 3: Comparison: Placebo vs Tio R1.25; Tio R1.25 minus Placebo; Test type: Superiority or Other; p = 0.0664, Mixed effect repeated measures (MMRM) — This test is considered as descriptive; This MMRM model includes treatment, period and baseline as fixed effects, and patient as a random effect; Mean Difference (Final Values) = 0.067, 95% CI [-0.005 to 0.138], Standard Error of Mean 0.036
Statistical Analysis 4: Comparison: Tio R1.25 vs Tio R5; Tio R5 minus Tio R1.25; Test type: Superiority or Other; Mixed effect repeated measures (MMRM); This MMRM model includes treatment, period and baseline as fixed effects, and patient as a random effect; Mean Difference (Final Values) = 0.046, 95% CI [-0.031 to 0.124], Standard Error of Mean 0.039
Statistical Analysis 5: Comparison: Tio R2.5 vs Tio R5; Tio R5 minus Tio R2.5; Test type: Superiority or Other; Mixed effect repeated measures (MMRM); This MMRM model includes treatment, period and baseline as fixed effects, and patient as a random effect; Mean Difference (Final Values) = 0.056, 95% CI [-0.014 to 0.126], Standard Error of Mean 0.036
Statistical Analysis 6: Comparison: Tio R1.25 vs Tio R2.5; Tio R2.5 minus Tio R1.25; Test type: Superiority or Other; Mixed effect repeated measures (MMRM); This MMRM model includes treatment, period and baseline as fixed effects, and patient as a random effect; Mean Difference (Final Values) = -0.010, 95% CI [-0.088 to 0.069], Standard Error of Mean 0.040

2. Secondary Outcome: Trough FEV1 Response
Description: The trough FEV1 is defined as the pre-dose FEV1 measured just prior to the last administration of randomised treatment. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing FEV1 data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre | 0.292 (0.045) | 0.384 (0.045) | 0.353 (0.045) | 0.442 (0.045)

3. Secondary Outcome: FEV1 Area Under the Curve From 0 to 3 h (AUC0-3h) Response
Description: FEV1 (AUC0-3h) will be calculated as the area under the curve from 0 to 3hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing FEV1 data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre | 0.363 (0.045) | 0.455 (0.045) | 0.434 (0.045) | 0.497 (0.045)

4. Secondary Outcome: FEV1 Individual Measurements Response at Each Time-point
Description: Individual FEV1 measurements at each time-point ("personal best"). Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks (10 min pre-dose, 30 min, 1,2,3 hours post-dose)
Population: FAS with non-missing FEV1 data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre
  Timepoint -0:10 hr response | 0.292 (0.045) | 0.384 (0.045) | 0.353 (0.045) | 0.442 (0.045)
  Timepoint 0:30 hr response | 0.337 (0.047) | 0.456 (0.047) | 0.407 (0.047) | 0.486 (0.047)
  Timepoint 1:00 hr response | 0.353 (0.048) | 0.456 (0.048) | 0.416 (0.048) | 0.505 (0.047)
  Timepoint 2:00 hr response | 0.394 (0.047) | 0.467 (0.048) | 0.453 (0.047) | 0.501 (0.047)
  Timepoint 3:00 hr response | 0.396 (0.048) | 0.467 (0.048) | 0.489 (0.048) | 0.497 (0.047)

5. Secondary Outcome: Forced Vital Capacity (FVC) Peak (0-3h) Response
Description: The FVC peak (0-3h) response is determined at the end of the 4 week treatment period. This is the difference between the maximum FVC measured within the first 3 hours post dosing and the FVC baseline measurement. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing FVC data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre | 0.546 (0.049) | 0.554 (0.049) | 0.554 (0.048) | 0.548 (0.048)

6. Secondary Outcome: FVC Trough Response
Description: The trough FVC response is defined as the pre-dose FVC measured just prior to the last administration of randomised treatment. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing FVC data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre | 0.357 (0.047) | 0.375 (0.047) | 0.381 (0.047) | 0.400 (0.047)

7. Secondary Outcome: FVC Area Under the Curve From 0 to 3 h (AUC0-3h) Response
Description: FVC (AUC0-3h) will be calculated as the area under the curve from 0 to 3hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing FVC data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre | 0.413 (0.046) | 0.441 (0.046) | 0.417 (0.045) | 0.429 (0.045)

8. Secondary Outcome: FVC Individual Measurements at Each Time-point
Description: Individual FVC measurements at each time-point ("personal best"). Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks (10 min pre-dose, 30 min, 1,2,3 hours post-dose)
Population: FAS with non-missing FVC data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Litre
  Timepoint -0:10 hr response | 0.357 (0.047) | 0.375 (0.047) | 0.381 (0.047) | 0.400 (0.047)
  Timepoint 0:30 hr response | 0.397 (0.049) | 0.434 (0.049) | 0.394 (0.049) | 0.409 (0.049)
  Timepoint 1:00 hr response | 0.417 (0.049) | 0.443 (0.050) | 0.387 (0.049) | 0.448 (0.049)
  Timepoint 2:00 hr response | 0.429 (0.048) | 0.438 (0.048) | 0.444 (0.048) | 0.423 (0.048)
  Timepoint 3:00 hr response | 0.430 (0.048) | 0.461 (0.048) | 0.454 (0.048) | 0.456 (0.048)

9. Secondary Outcome: Forced Expiratory Flow (FEF) 25-75% Individual Measurements Response at Each Time Point
Description: FEF 25-75% is the mean forced expiratory flow between 25% and 75% of the FVC determined at the end of the 4-week treatment period. This is often referred to as the maximum midexpiratory flow. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks (10 min pre-dose, 30 min, 1,2,3 hours post-dose)
Population: FAS with non-missing FEF data
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 49 | 47 | 47 | 50
Litre
  Timepoint -0:10 hr response | 0.242 (0.081) | 0.533 (0.082) | 0.380 (0.082) | 0.566 (0.080)
  Timepoint 0:30 hr response | 0.268 (0.083) | 0.643 (0.084) | 0.513 (0.084) | 0.647 (0.082)
  Timepoint 1:00 hr response | 0.321 (0.087) | 0.655 (0.087) | 0.569 (0.087) | 0.641 (0.086)
  Timepoint 2:00 hr response | 0.357 (0.088) | 0.678 (0.089) | 0.607 (0.089) | 0.622 (0.087)
  Timepoint 3:00 hr response | 0.329 (0.083) | 0.662 (0.084) | 0.616 (0.084) | 0.620 (0.083)

10. Secondary Outcome: Mean Morning Peak Expiratory Flow (PEF) Response
Description: Mean morning PEF assessed by patients at home. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing morning PEF data
Measure: Least Squares Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 73 | 75 | 73 | 79
Litre/min | 7.267 (6.152) | 18.613 (6.118) | 23.185 (6.146) | 20.491 (6.031)

11. Secondary Outcome: Mean Evening PEF Response
Description: Mean evening PEF assessed by patients at home. Response was defined as the change from baseline. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing evening PEF data
Measure: Least Squares Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 73 | 74 | 75 | 79
Litre/min | -0.552 (6.098) | 5.985 (6.089) | 18.971 (6.043) | 16.565 (5.970)

12. Secondary Outcome: Change From Baseline in the Number of Puffs of Rescue Medication Per Day
Description: Mean number of inhalations (puffs) of unscheduled rescue salbutamol therapy during whole day. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and 4 weeks
Population: FAS with non-missing data for rescue medication
Measure: Least Squares Mean (Standard Error); unit: Puffs/day
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 73 | 73 | 73 | 79
Puffs/day | -0.412 (0.155) | -0.635 (0.156) | -0.521 (0.154) | -0.528 (0.151)

13. Secondary Outcome: Control of Asthma as Assessed by Asthma Control Questionnaire (ACQ)
Description: ACQ is a questionnaire consisting of a seven point Likert scale ranging from 0 to 6, whereby 0 represents good control and 6 represents poor control of asthma. The scale describes the frequency and severity of asthma symptoms. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: 4 weeks
Population: FAS with non-missing ACQ data
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 74 | 73 | 74 | 77
Units on a scale | 1.371 (0.078) | 1.189 (0.079) | 1.366 (0.078) | 1.287 (0.078)

14. Secondary Outcome: Change From Baseline in Mean Number of Nighttime Awakenings
Description: Mean number of nighttime awakenings due to asthma symptoms as assessed by patients eDiary incorporated in the AM3® device. Analysis adjusted for treatment, period, patient and baseline using a mixed model.
Time Frame: Baseline and last week of treatment (week 4)
Population: FAS with non-missing data for nighttime awakenings
Measure: Least Squares Mean (Standard Error); unit: Night awakenings per week
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Number analyzed (Participants) | 73 | 75 | 73 | 79
Night awakenings per week | -0.086 (0.030) | -0.027 (0.030) | -0.074 (0.030) | -0.066 (0.029)

ADVERSE EVENTS:
Time Frame: 4 weeks + 30 days if in last period
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/75 | 0/75 | 1/80
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/75 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Tio R1.25 (N=75) | Tio R2.5 (N=75) | Tio R5 (N=80)
H1N1 influenza (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.